CLINICAL TRIAL: NCT01727505
Title: Volume Guarantee Ventilation in Preterm Infants With Frequent Episodes of Hypoxemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Nelson Claure, Research Associate Professor of Pediatrics, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20120623
Record Dates: First submitted 2012-11-08; First posted 2012-11-16 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Episodic Hypoxemia in Mechanically Ventilated Preterm Infants
Keywords: hypoxemia; desaturation; mechanical ventilation; preterm infants; volume guarantee ventilation
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A: Conventional-Volume Guarantee (Active Comparator): This is a crossover study. Infants will be assigned to one of two sequences. Sequence A consists of a 24-hour period during which the infant receives conventional mechanical ventilation followed by a second 24 hour period during which the infant receives volume guarantee ventilation.
  Interventions: Device: Sequence A: Conventional-Volume Guarantee
- Sequence B: Volume Guarantee-Conventional (Active Comparator): This is a crossover study. Infants will be assigned to one of two sequences. Sequence B consists of a 24-hour period during which the infant receives volume guarantee ventilation followed by a second 24 hour period during which the infant receives conventional mechanical ventilation.
  Interventions: Device: Sequence B: Volume Guarantee-Conventional

INTERVENTIONS:
Device: Sequence A: Conventional-Volume Guarantee — This is a crossover study. Infants will be randomly assigned to one of two sequences.
  In sequence A, the infant will undergo a 24-hour period of conventional mechanical ventilation followed by a 24 hour period of volume guarantee ventilation.
  Both conventional mechanical ventilation and volume guarantee ventilation will be provided by the same neonatal ventilator (AVEA, CareFusion Inc, Yorba Linda, CA).
  During the 24 hour period of conventional mechanical ventilation, the infant will receive mechanical ventilation with the settings determined by the clinical team.
  During volume guarantee ventilation, the set tidal volume to be maintained by the ventilator will be the average tidal volume delivered by the ventilator prior to start of study.
  Arms: Sequence A: Conventional-Volume Guarantee
Device: Sequence B: Volume Guarantee-Conventional — This is a crossover study. Infants will be randomly assigned to one of two sequences.
  In sequence B, the infant will undergo a 24-hour period of volume guarantee ventilation followed by a 24 hour period of conventional mechanical ventilation.
  Both conventional mechanical ventilation and volume guarantee ventilation will be provided by the same neonatal ventilator (AVEA, CareFusion Inc, Yorba Linda, CA).
  During the 24 hour period of conventional mechanical ventilation, the infant will receive mechanical ventilation with the settings determined by the clinical team.
  During volume guarantee ventilation, the set tidal volume to be maintained by the ventilator will be the average tidal volume delivered by the ventilator prior to start of study.
  Arms: Sequence B: Volume Guarantee-Conventional

SUMMARY:
Preterm infants undergoing mechanical ventilation often present with respiratory instability which leads to fluctuations in ventilation and oxygenation. In conventional modes of mechanical ventilation used in these patients, the ventilator delivers breaths at a set rate and a constant peak inspiratory pressure.

We have demonstrated that spontaneous episodes of hypoxemia in mechanically ventilated preterm infants are frequently triggered by a loss in end-expiratory lung volume followed by decrease in tidal volume. This is due to a reduction in respiratory system compliance and increase in airway resistance.

Volume Guarantee ventilation is a mode of ventilation in which ventilator measures the exhaled tidal volume of each ventilator breath and automatically adjusts the peak inspiratory pressure to deliver the set tidal volume. We have previously shown that Volume Guarantee reduced the severity and duration of hypoxemia episodes during a period of 2 hours in preterm infants The study hypothesis is that Volume Guarantee ventilation will decrease the duration of episodes of hypoxemia when compared to conventional mechanical ventilation during routine clinical conditions and over longer periods of time.

The objective of the study is to evaluate the effects of Volume Guarantee on the duration, severity and frequency of episodes of hypoxemia in mechanically ventilated preterm infants who present with frequent hypoxemia episodes in comparison to conventional ventilation over two periods of 24 hours each and under routine clinical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Born at less than 32 weeks of gestational age.
* Requiring mechanical ventilation on a mandatory ventilator rate greater than or equal to 20 per minute and receiving a mean tidal volume of at least 4 ml/kg.
* Presenting with 4 or more episodes of hypoxemia, defined as oxygen saturation less than 75%, in the 8 hours prior to the study.

Exclusion Criteria:

* Major congenital anomalies.
* Hemodynamic instability requiring inotropes within 72 hours prior to the study
* Culture proven sepsis within 72 hours prior to the study.
* Diagnosis of pulmonary interstitial emphysema or pneumothorax within the 72 hours prior to the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Claure, M.Sc., Ph.D., Principal Investigator — University of Miami; Eduardo Bancalari, M.D., Principal Investigator — University of Miami
Locations (1):
- Newborn Intensitve Care Unit at Holtz Children's Hospital of Jackson Health System, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the Project NewBorn Neonatal Intensive Care Unit of the Jackson Memorial Hospital/University of Miami Medical Center. Subjects were recruited into the study between December, 2012 and September, 2014.
Pre-assignment Details: 42 infants were screened. Of these, 9 declined participation and 3 did not meet inclusion criteria.
  30 infants were enrolled (consented). Of these, 4 infants became ineligible after consent and were not studied.
  26 enrolled infants were studied.
Groups:
- Sequence A: Conventional-Volume Guarantee: This is a crossover study. Each patient is randomly assigned to one of two sequences.
  Sequence A consisted of a 24-hour period during which the infant received conventional mechanical ventilation followed by a 24 hour period during which the infant received volume guarantee ventilation.
- Sequence B: Volume Guarantee-Conventional: This is a crossover study. Each patient is randomly assigned to one of two sequences.
  Sequence B consisted of a 24-hour period during which the infant received volume guarantee ventilation followed by a 24 hour period during which the infant received conventional mechanical ventilation.
Period: First 24 Hours
Arm/Group | Sequence A: Conventional-Volume Guarantee | Sequence B: Volume Guarantee-Conventional
Started | 14 | 12
Completed | 14 | 11
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second 24 Hours
Arm/Group | Sequence A: Conventional-Volume Guarantee | Sequence B: Volume Guarantee-Conventional
Started | 14 | 11
Completed | 14 | 10
Not Completed | 0 | 1
Not completed — Missing data | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Population: This is a crossover study. Infants were randomly assigned to one of two sequences.
  Sequence A consisted of 24 hours of Conventional Mechanical Ventilation followed by 24 hours of Volume Guarantee Ventilation.
  Sequence B consisted of 24 hours of Volume Guarantee Ventilation followed by 24 hours of Conventional Mechanical Ventilation.
Arm/Group | Study Population
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: days] | 32 (22)
Gender [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Gestational age [Mean (Standard Deviation); unit: weeks] | 25 (1.5)
Birth weight [Mean (Standard Deviation); unit: grams] | 685 (216)
Ventilator mandatory rate [Mean (Standard Deviation); unit: breaths per minute] | 33 (8.7)
Peak inspiratory pressure [Mean (Standard Deviation); unit: cm H2O] | 19.4 (1.5)
Pressure support [Mean (Standard Deviation); unit: cm H2O] | 10.4 (1.7)
Positive end expiratory pressure [Mean (Standard Deviation); unit: cm H2O] | 5.3 (0.47)
Fraction of Inspired Oxygen [Mean (Standard Deviation); unit: fraction] | 0.38 (0.09)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Spent With Arterial Oxygen Saturation < 75%
Description: Percentage of time spent with arterial oxygen saturation < 75%
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: % of time
Groups:
- Conventional Mechanical Ventilation Period; Volume Guarantee Ventilation Period: This is a crossover study that consisted of a 24-hour period during which the infant received conventional mechanical ventilation and another 24 hour period during which the infant received volume guarantee ventilation.
  The sequence of conventional and volume guarantee ventilation were assigned at random.
Arm/Group | Conventional Mechanical Ventilation Period | Volume Guarantee Ventilation Period
Number analyzed (Participants) | 24 | 24
% of time | 5 [3.9 to 6.9] | 4.4 [2.9 to 5]
Statistical Analysis 1: Comparison: Conventional Mechanical Ventilation Period vs Volume Guarantee Ventilation Period; Test type: Superiority or Other; p = 0.44, Wilcoxon signed rank test

2. Secondary Outcome: Frequency of Severe Hypoxemia Episodes
Description: Frequency of severe hypoxemia episodes defined as periods with arterial oxygen saturation SpO2 < 75% lasting for at least 20 seconds.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: severe hypoxemia episodes per hour
Arm/Group | Conventional Mechanical Ventilation Period | Volume Guarantee Ventilation Period
Number analyzed (Participants) | 24 | 24
severe hypoxemia episodes per hour | 2.1 [1.3 to 2.6] | 1.9 [1.1 to 2.5]
Statistical Analysis 1: Comparison: Conventional Mechanical Ventilation Period vs Volume Guarantee Ventilation Period; Test type: Superiority or Other; p = .75, Wilcoxon signed rank test

3. Secondary Outcome: Frequency of Hypoxemia Episodes
Description: Frequency of hypoxemia episodes defined as episodes with arterial saturation < 85% for at least 20 seconds
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: hypoxemia episodes per hour
Arm/Group | Conventional Mechanical Ventilation Period | Volume Guarantee Ventilation Period
Number analyzed (Participants) | 24 | 24
hypoxemia episodes per hour | 6.8 [4.6 to 7.9] | 6.5 [5.6 to 8.9]
Statistical Analysis 1: Comparison: Conventional Mechanical Ventilation Period vs Volume Guarantee Ventilation Period; Test type: Superiority or Other; p = 0.2, Wilcoxon signed rank test

4. Secondary Outcome: Duration of Hypoxemia Episodes
Description: Duration of hypoxemia episodes of arterial saturation < 85% for at least 20 seconds. Calculated as the mean episode duration per subject per period. Reported as median and inter-quartile range of all subjects.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Conventional Mechanical Ventilation Period | Volume Guarantee Ventilation Period
Number analyzed (Participants) | 24 | 24
seconds | 76 [70 to 92] | 73 [65 to 81]
Statistical Analysis 1: Comparison: Conventional Mechanical Ventilation Period vs Volume Guarantee Ventilation Period; Test type: Superiority or Other; p = 0.02, Wilcoxon signed rank test

5. Other Pre Specified Outcome: Fraction of Inspired Oxygen (FiO2)
Description: Calculated as the mean value of the recorded fraction of inspired oxygen for each subject during each of the two 24 hour periods.
  Reported as median and inter-quartile range of all subjects.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: fraction
Arm/Group | Conventional Mechanical Ventilation Period | Volume Guarantee Ventilation Period
Number analyzed (Participants) | 24 | 24
fraction | .42 [.37 to .53] | .41 [.36 to .46]
Statistical Analysis 1: Comparison: Conventional Mechanical Ventilation Period vs Volume Guarantee Ventilation Period; Test type: Superiority or Other; p = .049, Wilcoxon signed rank test

6. Other Pre Specified Outcome: Tidal Volume
Description: The mean exhaled tidal volume of mechanical breaths.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ml/Kg
Arm/Group | Conventional Mechanical Ventilation Period | Volume Guarantee Ventilation Period
Number analyzed (Participants) | 24 | 24
ml/Kg | 6.2 (1.6) | 5.6 (0.7)
Statistical Analysis 1: Comparison: Conventional Mechanical Ventilation Period vs Volume Guarantee Ventilation Period; Test type: Superiority or Other; p = 0.006, Paired t-test

ADVERSE EVENTS:
Groups:
- Conventional Mechanical Ventilation Period: This is a crossover study. Infants were randomly assigned to one of two sequences that consisted of a 24-hour period during which the infant received conventional mechanical ventilation and another 24 hour period during which the infant received volume guarantee ventilation.
  These data represent the 24 hours of Conventional Mechanical Ventilation.
- Volume Guarantee Ventilation Period: This is a crossover study. Infants were randomly assigned to one of two sequences that consisted of a 24-hour period during which the infant received conventional mechanical ventilation and another 24 hour period during which the infant received volume guarantee ventilation.
  These data represent the 24 hours of Volume Guarantee Ventilation.
Arm/Group | Conventional Mechanical Ventilation Period | Volume Guarantee Ventilation Period
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Mechanical Ventilation Period (N=25) | Volume Guarantee Ventilation Period (N=26)
Increased PaCO2 requiring high frequency ventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No